CLINICAL TRIAL: NCT06962163
Title: Prospective Phase 0 Pilot Study, Assessing Potential Interest of [68Ga]Ga-PentixaFor PET/CT in Metastatic Triple Negative Breast Cancer Patients
Brief Title: Assessement of Potential Interest of [68Ga]Ga-PentixaFor PET/CT in Metastatic Triple Negative Breast Cancer Patients
Acronym: EXIGENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-2023-17
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Triple negative breast cancer; [68Ga]Ga-PentixaFor PET/CT; [18F]FDG PET/CT; CXCR4
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: [68Ga]Ga-PentixaFor PET-CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-PentixaFor (Experimental): 2 [68Ga]Ga-PentixaFor PET-CT are performed after patient inclusion and at disease progression.
  Interventions: Diagnostic Test: [68Ga]Ga-PentixaFor PET/CT

INTERVENTIONS:
Diagnostic Test: [68Ga]Ga-PentixaFor PET/CT — [68Ga]Ga-PentixaFor PET-CT is performed after patient inclusion. The patient is treated as per standard of care until disease progression. Then another [68Ga]Ga-PentixaFor PET-CT is performed.

SUMMARY:
Triple-negative breast cancer (TNBC) is a particularly aggressive type of breast cancer that is difficult to treat. Unlike other forms of breast cancer, TNBC tends to relapse earlier and spread more quickly to other parts of the body. Unfortunately, patients with TNBC have a lower survival rate, often less than five years after diagnosis. This highlights the urgent need for better treatments for TNBC.

One of the main challenges in treating TNBC is that it lacks certain receptors that other breast cancers have. These receptors are usually targeted by specific therapies, making TNBC harder to treat with targeted approaches.

Currently, a type of imaging called [18F]FDG PET/CT is the most accurate method for detecting breast cancer and its spread. However, with the rise of personalized medicine, there is a growing interest in molecular targeted approaches. These methods aim to provide highly specific diagnostics and treatments based on the unique characteristics of each patient's cancer.

One promising target for these new approaches is a receptor called CXCR4. CXCR4 is found on the surface of many cells and is involved in various processes in the body. It is often overexpressed in different types of cancer, including breast cancer. Research has shown that CXCR4 levels are higher in metastatic sites (where cancer has spread) compared to primary tumors. CXCR4 is not only present in cancer cells but also in immune cells within the tumor environment.

In invasive breast cancer, CXCR4 plays a crucial role in tumor migration, invasiveness, metastasis, and proliferation. A clinical study evaluated 18 breast cancer patients using a new imaging method called [68Ga]Ga-PentixaFor PET/CT or PET/MR. They found that this method showed higher uptake in breast cancer cases with poorer prognosis compared to the traditional [18F]FDG PET/CT. Higher CXCR4 expression is particularly seen in TNBC compared to other breast cancer subtypes.

The goal of the study is to assess how [68Ga]Ga-PentixaFor is distributed in the body using PET/CT imaging. This will help demonstrate the potential of CXCR4 as a promising target for new treatments. If successful, [68Ga]Ga-PentixaFor PET/CT could become a valuable tool for identifying patients who might benefit from treatments using [177Lu]/[90Y] PentixaTher.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) is the most aggressive and hard-to-treat form of breast cancer. TNBC has a higher propensity for earlier relapse and an increased risk of metastasis than all other forms of breast cancer. TNBC patients have a low survival rate (<5 years). This clearly shows an urgent unmet medical need for TNBC patients. The lack of receptors makes it challenging to develop more effective targeted therapy to treat TNBC.

Currently, [18F]FDG PET/CT offer highest diagnostic accuracy in the detection of breast cancer and distant metastases. With the increasing role of personalized medicine, however, the desire for molecular targeted approaches emerged, enabling high-specificity diagnostics and molecular targeted therapies with the appropriate molecular key target.

CXCR4 is a 7-transmembrane G-coupled receptor belonging to the chemokine receptor family and is expressed by a variety of cells during development and thereafter. CXCR4 has been found to be overexpressed by various human cancers including breast cancer. The level of CXCR4 expression was shown to be higher in metastatic sites as compared to the primary tumours, and changes in CXCR4 signalling have been shown to significantly alter metastatic burden in animal models. CXCR4 is not only expressed by cancer cells themselves, but also by tumour-infiltrating immune cells. Within the tumour microenvironment, the major CXCR4-expressing cells are B-lymphocytes and plasmacytoid dendritic cells, both potentially contributing to an immunosuppressive site permissive for tumour progression.

CXCR4 is frequently overexpressed in invasive breast cancer and has an important role in tumour migration, invasiveness, metastasis, and proliferation (2).

Vag et al. evaluated 18 patients with breast cancer who underwent [68Ga]Ga-PentixaFor PET/CT or PET/MR (6). It was noted that a higher SUVmax of [18F]FDG was observed in all cases, compared with [68Ga]Ga-PentixaFor. It was also noted that the uptake seen in breast cancer is associated with a poorer prognosis. Higher CXCR4 expression is seen in triple-negative breast cancer compared to the luminal subtypes. [68Ga]Ga-PentixaFor PET/CT may have a role in prognostication of breast cancer.

The purpose of this trial is to assess the biodistribution of [68Ga]Ga-PentixaFor using PET/CT imaging, thus allowing us to demonstrate the potential of CXCR4 as a promising molecular target.

After establishing the targeting properties of [68Ga]Ga-PentixaFor PET/CT in TNBC, it could act as an effective companion imaging diagnostic and therefore a useful tool for identification of patients potentially benefiting from treatment using the theragnostic equivalent [177Lu]/[90Y] PentixaTher.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
2. Female or male, Age ≥ 18 years at time of study entry.
3. Primitive triple negative breast cancer proven histologically, defined according to the following criteria:

   * Estrogen receptors <10%.
   * And progesterone receptors <10%.
   * And HER2 not amplified or not overexpressed.
4. Recurrence metastatic Breast Cancer or De Novo metastatic Breast Cancer documented by [18F]FDG PET/CT ± conventional imaging with at least one measurable metastasis according to PERCIST and/or RECIST.
5. ECOG performance status < 2.
6. Negative serum/urine pregnancy test prior to [68Ga]Ga-PentixaFor administration for female patient of childbearing potential*.
7. Consent to use a contraception method for at least 3 months after each administration of [68Ga]Ga-PentixaFor (as defined in Appendix 7 and according to local guidelines).
8. Adequate Organ function confirmed by laboratory tests results allowing for safe administration of [68Ga]Ga- PentixaFor:

   Hematologic function: Absolute Neutrophil Count (ANC) of ≥ 1.5 x 109 /L, platelet count of ≥ 100 x 109 /L, and hemoglobin of ≥ 9 g/dL).

   Hepatic function: AST and ALT ≤ 3 x ULN (≤ 5 x ULN if liver metastases).
9. Renal function: Estimated Glomerular Filtration Rate (eGFR) ≥ 50 mL/min/1.73m², as calculated using the CKD-EPI or MDRD equation.Life expectancy at least 3 months.
10. Patient has valid health insurance.
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

    * Note: a female participant of childbearing potential is a woman who is not permanently sterilized or not postmenopausal (postmenopausal is defined as 12 months with no menses without an alternative medical cause).

Exclusion Criteria:

1. History of another primary malignancy within the last 3 years before study entry except for basal cell carcinoma.
2. Impossibility to hold lying motionless at least 1 hour, or known claustrophobia.
3. Serious non-malignant disease (e.g. psychiatric, infectious, autoimmune or metabolic), that may interfere with the objectives of the study or with the safety or compliance of the subject, as judged by the investigator.
4. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
5. Pregnant, likely to be pregnant or breastfeeding woman.
6. Blood glucose > 12mmol/L.
7. Renal insufficiency with GFR ≤ 45 mL/min/ 1.73 m².
8. Known hypersensitivity to any active pharmaceutical agent or constituent of the [68Ga]Ga-PentixaFor and/or [18F]FDG product.
9. Body weight of less than 48 kg.
10. Persons deprived of their liberty, under a measure of safeguard of justice, under guardianship or placed under the authority of a guardian.
11. Disorder precluding understanding of trial information or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
To assess the concordance for tumour lesion detection with [68Ga]Ga-PentixaFor PET/CT and [18F]FDG PET/CT based on a lesion-by-lesion basis analysis performed at patient inclusion | 1 day
  Concordance study of metastatic uptake seen in [18F]FDG PET/CT scan and [68Ga]Ga-PentixaFor PET/CT scan per "lesion" by comparing for each lesion the [18F]FDG PET scan and [68Ga]Ga-PentixaFor PET/CT scan by assessing a ratio "Number of positive or negative [68Ga]Ga-PentixaFor lesions / Number of positive or negative FDG lesions" performed at patient inclusion

SECONDARY OUTCOMES:
To assess the concordance for tumour lesion detection with [68Ga]Ga-PentixaFor PET/CT and [18F]FDG PET/CT based on a lesion-by-lesion basis analysis performed at disease progression | 36 months
  Concordance study of metastatic uptake seen in [18F]FDG PET/CT scan and [68Ga]Ga-PentixaFor PET/CT scan per "lesion" by comparing for each lesion the [18F]FDG PET/CT scan and [68Ga]Ga-PentixaFor PET/CT scan by assessing a ratio "Number of positive or negative [68Ga]Ga-PentixaFor lesions / Number of positive or negative FDG lesions" performed at disease progression
To assess the concordance for tumour lesion detection with [68Ga]Ga-PentixaFor PET/CT and conventional imaging CT scan based on a lesion-by-lesion basis analysis performed at patient inclusion | 1 day
  Conventional imaging (CT scan), and [68Ga]Ga-PentixaFor PET/CT will be analysed for each lesion, obtaining a ratio of number of [68Ga]Ga-PentixaFor(+) lesions / number of CT scan lesions" at patient inclusion
To assess the concordance for tumour lesion detection with [68Ga]Ga-PentixaFor PET/CT and conventional imaging: CT scan based on a lesion-by-lesion basis analysis performed at disease progression | 36 months
  Conventional imaging: CT scan, and [68Ga]Ga-PentixaFor PET/CT will be analysed for each lesion, obtaining a ratio of number of [68Ga]Ga-PentixaFor(+) lesions / number of CT scan lesions" at disease progression
To determine the percentage of total tumour burden (whole body) detected on [68Ga]Ga-PentixaFor PET/CT compared to that defined on [18F]FDG PET/CT (considered as reference). | 36 months
  Percentage of [68Ga]Ga-PentixaFor(+) metastatic tumour burden compared to total metastatic tumour burden by [18F]FDG PET/CT
To assess the correlation between the standard uptake values (SUV) of [68Ga]Ga-PentixaFor and CXCR4 expression by IHC assessment on primitive and/or metastatic tumour samples at screening and at disease progression if a biopsy is performed | 36 months
  Assess the correlation between the standard uptake values (SUV) of [68Ga]Ga-PentixaFor and IHC CXCR4 expression, by comparing the [68Ga]Ga-PentixaFor semi-quantitative data with the CXCR4 expression results of biopsied metastases at screening and at disease progression if biopsy is performed
To assess the safety and tolerance of [68Ga]Ga-PentixaFor | 2 days
  The tolerance of [68Ga]Ga-PentixaFor will be checked by measuring and monitoring vital signs for 60 minutes after [68Ga]Ga-PentixaFor administration. The patient will be informed that in the event of abnormal physical signs, occurring within 48 hours after [68Ga]Ga-PentixaFor administration, he (she) must inform the investigator for registration. The CTC-NCI Common Toxicity Criteria, version 5.0 reference will be used

OTHER OUTCOMES:
To assess the prognostic value of serum FLT3-Ligand in relapsing Triple Negative Breast Cancer patients | 36 months
  Plasma FLT3-Ligand dosage will be performed at screening, every 3 months during treatment period and at disease progression follow-up visit for all patients.
  The relationship between FLT3-Ligand levels and patient outcomes (OS and DFS) will be analysed using Kaplan-Meier survival analysis and univariable Cox analysis

CONTACTS AND LOCATIONS:
Overall Officials: CAROLINE ROUSSEAU, MD, PhD, Principal Investigator — Institut de Cancérologie de l'Ouest (ICO)
Locations (1):
- Institut de cancerologie de l'Ouest, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No
The IPD data is confidential.